CLINICAL TRIAL: NCT06569602
Title: Edwards EVOQUE Transcatheter Tricuspid Valve Replacement: Real World European Investigation of Safety and Clinical Efficacy Using a Novel Device
Brief Title: Real World European Investigation of Safety and Clinical Efficacy of the EVOQUE System (TRISCEND III EU)
Status: Recruiting | Type: Observational
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: 2024-07
Record Dates: First submitted 2024-08-12; First posted 2024-08-26 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Tricuspid Valve Regurgitation; Heart Valve Diseases; Cardiovascular Diseases
MeSH Terms: conditions — Tricuspid Valve Insufficiency; Heart Valve Diseases; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Treatment: Treatment with the Edwards EVOQUE Tricuspid Transcatheter Valve Replacement System
  Interventions: Device: Transcatheter Tricuspid Valve Replacement

INTERVENTIONS:
Device: Transcatheter Tricuspid Valve Replacement — Replacement of the tricuspid valve through a transcatheter approach
  Other Names: Edwards EVOQUE Tricuspid Valve Replacement System

SUMMARY:
This is a prospective, single-arm, multi-center, real-world study of an the Edwards EVOQUE system.

DETAILED DESCRIPTION:
This is a prospective, single-arm, multi-center, real-world study of an approved device. Up to 500 patients will be enrolled in this study at up to 45 sites in Europe. All enrolled patients will be assessed at the following intervals: baseline, index procedure, discharge (or 7-days post-index procedure whichever occurs first), 30 days, 1 year, and annually through 5 years.

Study enrollment is expected to last approximately 2-4 years, followed by 5 years of follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. The Local Site Heart Team determines that the patient is appropriate for transcatheter tricuspid valve replacement with the EVOQUE system per the current instructions for use.
2. Patient agrees to attend follow-up assessments.
3. Patients provided written informed consent for participation in the study.

Exclusion Criteria:

1. Patient participating in another interventional biologic, drug, or device clinical study that has not met its primary endpoint(s).
2. Any patient considered to be part of a vulnerable population.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with at least severe tricuspid regurgitation who are candidates for transcatheter tricuspid valve replacement, selected to receive treatment with the EVOQUE system per the current Instructions for use, and meet the eligibility requirements.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2030-09-30 (Estimated); Study Completion 2033-09-30 (Estimated)

PRIMARY OUTCOMES:
Tricuspid regurgitation grade | Up to 7 days, 30 days, and 1 year
  Number of patients with optimal TR grade (≤1 on a 0-5 grade scale)
Number of patients with major adverse events (MAE rates) | 30 days
  The primary safety endpoint is the proportion of patients with major adverse events (MAEs) at 30 days

SECONDARY OUTCOMES:
All-cause mortality | 30 days, 1 year, and 2 years
  Number of participants with all-cause mortality
Cardiovascular mortality | 30 days, 1 year, and 2 years
  Number of participants with cardiovascular mortality
Heart failure hospitalizations | 30 days, 1 year, and 2 years
  Number of patients with heart failure hospitalizations
Tricuspid valve re-intervention | 30 days, 1 year, and 2 years
  Number of participants with tricuspid valve re-intervention
Health Status - Assessed by Kansas City Cardiomyopathy Questionaire (KCCQ) Scores | 30 days, 1 year, and 2 years
  KCCQ is a 23-item, self-administered, validated questionnaire that quantifies physical function, symptoms, social function, self-efficacy, and quality of life for patients with heart failure. Scores range from 0 to 100 with higher scores indicating better function (100 = no symptoms, no limitations, and excellent quality of life).
NYHA Functional Class | 30 days, 1 year, and 2 years
  Number of patients with improvement in NYHA class

CONTACTS AND LOCATIONS:
Overall Officials: Volker Rudolph, Prof. MD, Principal Investigator — Herz-und Diabeteszentrum NRW, Bad Oeynhausen; Fabien Praz, Prof. MD, Principal Investigator — Bern, Insespital, Switzerland
Locations (2):
- Herz-und Diabeteszentrum NRW, Bad Oeynhausen, Germany
- Inselspital, Bern, Switzerland